CLINICAL TRIAL: NCT02876133
Title: Improving Colorectal Cancer Screening: Using Narrow Band Imaging for Colonic Sessile Serrated Lesions
Brief Title: Narrow Band Imaging Versus White Light for Colonoscopy Serrate Lesions Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Beatriz Ângelo (Other)
Responsible Party: Principal Investigator, Alexandre Ferreira, Gastroenterologist, Hospital Beatriz Ângelo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 176
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Colon Cancer; Colon Sessile Serrated Adenoma/Polyp
MeSH Terms: conditions — Colonic Neoplasms; Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narrow band imaging withdrawal (Experimental): colonoscope withdrawal and mucosal inspection performed under narrow band imaging
  Interventions: Device: narrow band imaging withdrawal
- white light withdrawal (Placebo Comparator): colonoscope withdrawal and mucosal inspection performed under white light imaging
  Interventions: Device: white light withdrawal

INTERVENTIONS:
Device: narrow band imaging withdrawal — colonoscope withdrawal and mucosal inspection performed under narrow band imaging
  Arms: Narrow band imaging withdrawal
Device: white light withdrawal — colonoscope withdrawal and mucosal inspection performed under white light imaging
  Arms: white light withdrawal

SUMMARY:
Colorectal cancer (CRC) is a leading cause of cancer death and its' incidence is rising in most European countries. Colonoscopy has been shown to reduce CRC incidence, however its effectiveness depends on the sensitivity to detect pre-malignant lesions.

Our aim is to evaluate narrow band imaging (NBI) during colonoscopy and serum miRNAs as novel tools for the early detection of colonic sessile serrated lesions (SSL). The investigators will perform a multicenter-randomized-controlled-trial to study the role of NBI in SSL detection.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective colonoscopies

Exclusion Criteria:

* known polyposis syndromes
* primary sclerosing cholangitis
* inflammatory bowel disease
* personal colorectal cancer history

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 987 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
average number of serrated lesions ≥10 mm detected per colonoscopy | immediate

SECONDARY OUTCOMES:
Serrated class lesions detection rate | immediate
  number of patients with at least 1 lesion/total number of participants
Serrated lesions <10 mm detected per colonoscopy | immediate
SSL detection rate | immediate
  histologically defined according to the WHO criteria
Adenoma detection rate | immediate
  number of patients with at least 1 adenoma/total number of participants
Adenomas detected per colonoscopy | immediate
Advanced (malignant) adenocarcinoma detection rate | immediate
Incidence of procedure related adverse events | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre O Ferreira, MD, Principal Investigator — Hospital Beatriz Ângelo
Locations (3):
- Portugal (3):
  - Hospital Beatriz Ângelo, Loures
  - Centro Hospitalar do Porto, Porto
  - Instituto Português de Oncologia do Porto, Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK, Ahnen DJ, Baron JA, Batts KP, Burke CA, Burt RW, Goldblum JR, Guillem JG, Kahi CJ, Kalady MF, O'Brien MJ, Odze RD, Ogino S, Parry S, Snover DC, Torlakovic EE, Wise PE, Young J, Church J. Serrated lesions of the colorectum: review and recommendations from an expert panel. Am J Gastroenterol. 2012 Sep;107(9):1315-29; quiz 1314, 1330. doi: 10.1038/ajg.2012.161. Epub 2012 Jun 19. PMID 22710576